CLINICAL TRIAL: NCT04151667
Title: Phase II Study of Daratumumab Based Response Adapted Therapy for Older Adults With Newly Diagnosed Multiple Myeloma
Brief Title: Daratumumab Based Response Adapted Therapy for Older Adults With Newly Diagnosed Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20130
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Results first posted 2024-12-30 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
Keywords: myeloma; daratumumab
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — daratumumab; Dexamethasone; Calcium Dobesilate; Lenalidomide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- A: Daratumumab & Dexamethasone (Experimental): All participants will receive 1800 mg in 15 ml Daratumumab by subcutaneous injection weekly and be given 20 mg of Dexamethasone orally once a week for 2 months. Patients who receive a partial response or better will continue on this arm.
  Interventions: Drug: Daratumumab Injection; Drug: Dexamethasone Oral
- B: Daratumumab, Dexamethasone and Lenalidomide (Experimental): Participants who have less than a partial response to Arm A may have Lenalidomide added to their treatment. Lenalidomide will be given orally on days 1-21 of each 28 day treatment cycle.
  Interventions: Drug: Daratumumab Injection; Drug: Dexamethasone Oral; Drug: Lenalidomide Pill
- C: Daratumumab, Dexamethasone and Bortezomib (Experimental): Participants who have less than a partial response to Arm A may have Bortezomib added to their treatment. Bortezomib will be given weekly in subcutaneous injections at a starting dose of 1/3 mg/m^2 Days 1,8 and 15 of each 28 day treatment cycle.
  Interventions: Drug: Daratumumab Injection; Drug: Dexamethasone Oral; Drug: Bortezomib Injection

INTERVENTIONS:
Drug: Daratumumab Injection — Patient will receive daratumumab (1800 mg in 15 ml) administered by manual subcutaneous injections weekly for the first 8 weeks, every other week for the next 16 weeks and every 4 weeks after.
  Other Names: Darzalex
Drug: Dexamethasone Oral — The dexamethasone starting dose will be 20 mg PO once a week. Commercial dexamethasone will be used. Dexamethasone is often supplied in 4 mg tablets. Accordingly, patients will take 5 (4 mg tablets) one day of the week prior to the administration of daratumumab if this corresponds to a daratumumab dosing days. In non daratumumab dosing days, dexamethasone will be taken by the patient at home, usually in the morning with breakfast.
  Other Names: Decadron
Drug: Lenalidomide Pill — Lenalidomide will be given orally on days 1-21 of a 28 days cycle. The starting dose of lenalidomide will be based on the patient creatinine clearance per the package insert.
  Specifically patients with a creatinine clearance ≥ 50 ml/min will receive 25 mg of lenalidomide PO Days 1-21. Patients with a creatinine clearance ≥ 30 but less than 50 ml/min will receive 10 mg of lenalidomide.
  Patients with a creatinine clearance < 30 ml/min are not eligible but patients who experience a deterioration in the renal function during screening or treatment may continue on lenalidomide therapy as long as the risk / benefit profile is deemed acceptable, that study therapy is in the best interest of the patient and after discussion with the study principal investigator / sponsor.
  Other Names: Revlimid
  Arms: B: Daratumumab, Dexamethasone and Lenalidomide
Drug: Bortezomib Injection — Bortezomib will be given weekly subcutaneously in an effort to decrease the toxicity of the therapy. Specifically patients will receive a starting dose of bortezomib of 1.3 mg/m^2 Days 1,8,15 of a 28 day cycle. Bortezomib will be administered in the cancer center per standard of care procedures.
  Other Names: Velcade
  Arms: C: Daratumumab, Dexamethasone and Bortezomib

SUMMARY:
This is a Phase II study of daratumumab based therapies for older adults with multiple myeloma.

DETAILED DESCRIPTION:
In this response adapted approach, older adults with newly diagnosed symptomatic multiple myeloma will receive daratumumab and dexamethasone for 2 months. Patients who achieve a partial response or better will continue on daratumumab. Patients who achieve less than a partial response will have lenalidomide or bortezomib added to their therapy. Patients who experience progressive disease on daratumumab after the initial 2 months of monotherapy or on the combination of daratumumab and either lenalidomide or bortezomib will come off study

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Age 65 years or older and presence of coexisting conditions which in the opinion of the treating physician are likely to result in the development of unacceptable side effects associated with high-dose chemotherapy with stem-cell transplantation
* Able to adhere to the study visit schedule and other protocol requirements.
* Diagnosed with multiple myeloma and be considered to have active disease with either elevated Calcium, Renal Failure, Anemia, Bone Lesions (CRAB) criteria (hypercalcemia, renal failure, anemia, or bone lesions) or myeloma defining events (bone marrow ≥ 60% plasma cells, serum free light chain (sFLC) ratio≥ 100 or MRI or Positron Emission Tomography [PET] defined lesions). Patients must not have received an active chemotherapy regimen. Patients may have received palliative radiotherapy at least 2 weeks prior to the study start. Dexamethasone up to 160 mg total dose is allowed prior to participation
* Measurable myeloma paraprotein levels in serum (≥ 0.5 g/dL), urine (≥ 0.2 g excreted in a 24-hour urine collection sample) or by serum free light chains (involved free light chain greater than 100mg/L)
* Eastern Cooperative Group (ECOG) Performance Status of 0 - 2.
* Serum bilirubin levels </=1.5 times the upper limit of the normal range for the laboratory (ULN).
* Serum Aspirtate Transaminase (AST) or serum Alanine Aminotransferase (ALT) levels </=2 x Upper Limit of Normal (ULN)
* Must have adequate bone marrow function: a. Absolute neutrophil count > 1,000 cells/mm3 (1.0 x 109/L). b. Platelets >/= 75,000 /mm3.
* Hemoglobin > 8 g/dL (transfusions are allowed)
* Calculated creatinine clearance >/=30ml/min by Cockcroft-Gault formula.
* Men must agree to use a latex condom during sexual contact with a female of child bearing potential even if they have had a successful vasectomy. See Appendix C: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.

Exclusion Criteria:

* Ongoing severe infection requiring intravenous antibiotic treatment.
* Prior malignancy, except for adequately treated basal cell or squamous cell skin cancer, in-situ cervical cancer, or other cancer from which the subject has been disease-free for at least 2 years.
* Solitary bone or solitary extramedullary plasmacytoma as the only evidence of plasma cell dyscrasia.
* Patients with known Chronic Obstructive Pulmonary Disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal and , moderate or severe persistent asthma within the past 2 years or uncontrolled asthma. Patients with a history of COPD will have pulmonary function testing to include FEV1
* Uncontrolled medical problems such as diabetes mellitus, congestive heart failure, coronary artery disease, hypertension, unstable angina, arrhythmias), pulmonary, hepatic and renal diseases unless renal insufficiency is felt to be secondary to multiple myeloma.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Concurrent use of other anti-cancer agents or treatments with the exception for hormonal therapy, which is allowed.
* Known allergy or hypersensitivity or intolerance to any of the study drugs, hyaluronidase, monoclonal antibodies (mAbs), human proteins, or their excipients (refer to daratumumab IB), or known sensitivity to mammalian derived products
* Seropositive for human immunodeficiency virus (HIV)
* Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
* Seropositive for hepatitis C (except in the setting of a Sustained Virologic Response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-11-22 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2026-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Rachid C Baz, MD, Principal Investigator — H. Lee Moffitt Cancer & Research Institute
Locations (1):
- H. Lee Moffitt Cancer & Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Meads MB, Zhao X, Noyes DR, Sudalagunta P, Achille A, Zhang C, Renatino Canevarolo R, Silva M, Magaletti D, DeAvila D, Toska S, Oates A, Lastorino D, Idiaquez DW, Song J, Sansil S, Yoder SJ, Grajales-Cruz AF, Blue BJ, Freeman CL, Kim J, Alsina M, Brayer J, Siqueira Silva A, Song X, Shain KH, Baz RC. Target antigen and plasma cell phenotype are critical factors for sensitivity to response-adapted daratumumab therapy. Blood. 2025 Sep 22:blood.2025029921. doi: 10.1182/blood.2025029921. Online ahead of print. PMID 40983035

RESULTS

PARTICIPANT FLOW:
Groups:
- B: Daratumumab, Dexamethasone and Lenalidomide: Participants who have less than a partial response to Arm A may have Lenalidomide added to their treatment. Lenalidomide will be given orally on days 1-21 of each 28 day treatment cycle.
  Daratumumab Injection: Patient will receive daratumumab (1800 mg in 15 ml) administered by manual subcutaneous injections weekly for the first 8 weeks, every other week for the next 16 weeks and every 4 weeks after.
  Dexamethasone Oral: The dexamethasone starting dose will be 20 mg PO once a week.
  Patients will take 5 (4 mg tablets) one day of the week prior to the administration of daratumumab if this corresponds to daratumumab dosing days.
  Non daratumumab dosing days, dexamethasone will be taken by the patient at home.
  Lenalidomide Pill: Lenalidomide will be given orally on days 1-21 of a 28 days cycle. The starting dose of lenalidomide will be based on the patient creatinine clearance per the package insert.
  Specifically patients with a creatinine clearance ≥ 50 ml/min will receive 25 mg of lenalidomide PO Days 1-21. Patients with a creatinine clearance ≥ 30 but less than 50 ml/min will receive 10 mg of lenalidomide.
  Patients with a creatinine clearance < 30 ml/min are not eligible. Patients who experience a deterioration in renal function during screening or treatment may continue on lenalidomide therapy as long as the risk / benefit profile is deemed acceptable after discussion with the study principal investigator / sponsor.
Period: Overall Study
Arm/Group | A: Daratumumab & Dexamethasone | B: Daratumumab, Dexamethasone and Lenalidomide | C: Daratumumab, Dexamethasone and Bortezomib
Started | 14 | 12 | 7
Completed | 14 | 12 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Evaluable Participants
Groups:
- B: Daratumumab, Dexamethasone and Lenalidomide: Participants who have less than a partial response to Arm A may have Lenalidomide added to their treatment. Lenalidomide will be given orally on days 1-21 of each 28 day treatment cycle.
  Daratumumab Injection: Patient will receive daratumumab (1800 mg in 15 ml) administered by manual subcutaneous injections weekly for the first 8 weeks, every other week for the next 16 weeks and every 4 weeks after.
  Dexamethasone Oral: The dexamethasone starting dose will be 20 mg PO once a week. Commercial dexamethasone will be used. Dexamethasone is often supplied in 4 mg tablets. Accordingly, patients will take 5 (4 mg tablets) one day of the week prior to the administration of daratumumab if this corresponds to a daratumumab dosing days. In non daratumumab dosing days, dexamethasone will be taken by the patient at home, usually in the morning with breakfast.
  Lenalidomide Pill: Lenalidomide will be given orally on days 1-21 of a 28 days cycle.
  Specifically patients with a creatinine clearance ≥ 50 ml/min will receive 25 mg of lenalidomide PO Days 1-21. Patients with a creatinine clearance ≥ 30 but less than 50 ml/min will receive 10 mg of lenalidomide.
  Patients with a creatinine clearance < 30 ml/min are not eligible but patients who experience a deterioration in the renal function during screening or treatment may continue on lenalidomide therapy as long as the risk / benefit profile is deemed acceptable.
- Total: Total of all reporting groups
Arm/Group | A: Daratumumab & Dexamethasone | B: Daratumumab, Dexamethasone and Lenalidomide | C: Daratumumab, Dexamethasone and Bortezomib | Total
Number analyzed (Participants) | 14 | 12 | 7 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 14 | 12 | 7 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 3 | 15
  Male | 10 | 4 | 4 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 3
  Not Hispanic or Latino | 14 | 10 | 5 | 29
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 5
  White | 12 | 10 | 5 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 7 | 33

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall Response Rate of the response adapted strategy using the uniform response criteria of the International Myeloma Working Group (IMWG).
  Stringent Complete Response (sCR): Below plus normal FLC ratio and absence of clonal cells in bone marrow3 by immunohistochemistry or immunofluorescence Complete Response (CR): Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow Very Good Partial Response (VGPR): Serum and urine M-protein detectable by immunofixation but not on electrophoresis or > 90% reduction in serum M-protein plus urine M-protein level < 100 mg/24 h Partial Response (PR): > 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or to < 200 mg/24 h Minimal Response (MR): 25%-49% reduction of serum M-protein and 50%-89% reduction in 24 hours urinary M-protein Stable Disease (SD): Not meeting criteria for sCR, CR, VGPR, PR, MR, or Progressive Disease (PD)
Time Frame: Up to 8 months
Population: Evaluable Participants
Measure: Count of Participants; unit: Participants
Arm/Group | A: Daratumumab & Dexamethasone | B: Daratumumab, Dexamethasone and Lenalidomide | C: Daratumumab, Dexamethasone and Bortezomib
Number analyzed (Participants) | 12 | 12 | 7
Participants
  Stringent Complete Response | 1 | 1 | 0
  Complete Response | 1 | 1 | 0
  Very Good Partial Response | 7 | 9 | 5
  Partial Response | 3 | 1 | 1
  Minimal Response | 0 | 0 | 0
  Stable Disease | 0 | 0 | 1
  Progressive Disease | 0 | 0 | 0
  Partial Response and Better | 12 | 12 | 6

2. Secondary Outcome: Progression Free Survival
Description: Progression Free Survival (PFS) from start of treatment to death of any cause, disease progression or relapse of the date of last follow-up, whichever comes first. he PFS will be estimated by the Kaplan-Meier method and 95% confidence interval (CI) will be computed by complementary log-log transformation. The 1 and 2 year PFS and 95% Confidence Intervals will be reported.
Time Frame: Up to 2 years
Reporting Status: Not Posted

3. Secondary Outcome: Overall Survival
Description: Overall Survival (OS) from start of treatment to death of any cause or the date of last follow-up, whichever comes first. OS will be estimated by the Kaplan-Meier method and 95% confidence interval will be computed by complementary log-log transformation. The 2 year OS and 95% CI will be reported.
Time Frame: Up to 2 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Number of Participants Who Continue on Arm A After 2 Cycles
Description: The number of participants who continue on Daratumumab and Dexamethasone after 2 cycles
Time Frame: At the end of Cycle 2 (each cycle is 28 days)
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Number of Participants Without Minimal Residual Disease
Description: The number of patients who are without minimal residual disease (MRD) using Next Generation Sequencing (NGS) will be estimated and the 95% confidence interval will be computed by the Clopper-Pearson method.
Time Frame: Up to 8 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events are still being collected. Per Protocol, Adverse Events are collected from "On Treatment" date to 30 days after "Off Treatment" date (on average of 2 years)
Arm/Group | A: Daratumumab & Dexamethasone | B: Daratumumab, Dexamethasone and Lenalidomide | C: Daratumumab, Dexamethasone and Bortezomib
All-Cause Mortality (participants affected / at risk) | 1/33 | 1/12 | 0/7
Serious Adverse Events (participants affected / at risk) | 4/33 | 6/12 | 2/7
Other Adverse Events (participants affected / at risk) | 31/33 | 12/12 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Daratumumab & Dexamethasone (N=33) | B: Daratumumab, Dexamethasone and Lenalidomide (N=12) | C: Daratumumab, Dexamethasone and Bortezomib (N=7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchial infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fracture (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — Suspected tuberculosis
Sinus bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Daratumumab & Dexamethasone (N=33) | B: Daratumumab, Dexamethasone and Lenalidomide (N=12) | C: Daratumumab, Dexamethasone and Bortezomib (N=7)
Investigations, Other (Investigations) | 20 (106) | 8 (51) | 6 (32)
Blood lactate dehydrogenase increased (Investigations) | 15 (33) | 5 (7) | 4 (11)
Lymphocyte count decreased (Investigations) | 6 (14) | 5 (13) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (10) | 7 (18) | 2 (3)
Alkaline phosphatase increased (Investigations) | 4 (5) | 6 (9) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 2 (2) | 4 (9) | 1 (2)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (13) | 2 (2)
Platelet count decreased (Investigations) | 3 (4) | 2 (2) | 2 (5)
Blood bilirubin increased (Investigations) | 2 (13) | 2 (8) | 0 (0)
Creatinine increased (Investigations) | 3 (4) | 1 (7) | 1 (2)
Weight gain (Investigations) | 2 (3) | 1 (2) | 1 (1)
Weight loss (Investigations) | 1 (1) | 3 (3) | 0 (0)
White blood cell decreased (Investigations) | 3 (6) | 1 (2) | 1 (1)
Hemoglobin increased (Investigations) | 0 (0) | 1 (6) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 17 (45) | 10 (27) | 3 (8)
Hyperkalemia (Metabolism and nutrition disorders) | 13 (19) | 6 (12) | 4 (7)
Hypokalemia (Metabolism and nutrition disorders) | 2 (7) | 8 (21) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 11 (18) | 6 (13) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 6 (11) | 2 (2) | 3 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (8) | 5 (11) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 7 (16) | 1 (4) | 3 (10)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (7) | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (4) | 3 (4) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (3) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (2) | 1 (3) | 0 (0)
Hyperlipidemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 8 (10) | 9 (41) | 1 (3)
Constipation (Gastrointestinal disorders) | 9 (10) | 5 (9) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 6 (6) | 4 (7) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (3) | 4 (7) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (6) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Esophageal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Esophageal stenosis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 8 (10) | 5 (8) | 2 (2)
Fatigue (General disorders) | 8 (13) | 5 (12) | 1 (2)
Pain (General disorders) | 7 (10) | 3 (5) | 2 (4)
Fever (Gastrointestinal disorders) | 2 (2) | 3 (9) | 2 (3)
Injection site reaction (General disorders) | 3 (3) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 0 (0) | 2 (2)
Flu like symptoms (General disorders) | 2 (3) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (4) | 1 (1) | 0 (0)
Localized edema (General disorders) | 1 (1) | 0 (0) | 1 (2)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 0 (0)
Generalized edema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 (23) | 5 (9) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (20) | 6 (14) | 2 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4 (7) | 4 (6) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 3 (6) | 3 (4) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (3) | 2 (3) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 8 (13) | 6 (13) | 3 (4)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (9) | 0 (0)
Bronchial infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Sinusitis (Infections and infestations) | 1 (5) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Prostate infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 1 (3) | 0 (0)
Shingles (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 8 (12) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 5 (11) | 3 (4)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 2 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 4 (7) | 5 (6) | 1 (1)
Headache (Nervous system disorders) | 2 (6) | 4 (9) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 1 (1) | 4 (13)
Paresthesia (Nervous system disorders) | 3 (4) | 2 (2) | 1 (1)
Tremor (Nervous system disorders) | 3 (3) | 2 (3) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 3 (8) | 0 (0)
Memory impairment (Nervous system disorders) | 2 (2) | 1 (2) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4) | 4 (8) | 3 (8)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (10) | 2 (6) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (4) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash acneiform (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 7 (12) | 7 (12) | 4 (5)
Bruising (Injury, poisoning and procedural complications) | 5 (5) | 4 (4) | 1 (3)
Fracture (Injury, poisoning and procedural complications) | 5 (7) | 4 (5) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Intraoperative musculoskeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (10) | 5 (9) | 2 (3)
Agitation (Psychiatric disorders) | 2 (4) | 3 (4) | 1 (4)
Confusion (Psychiatric disorders) | 1 (1) | 3 (6) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (4) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (2) | 2 (4) | 0 (0)
Irritability (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 6 (6) | 3 (3) | 3 (6)
Blurred vision (Eye disorders) | 2 (3) | 2 (2) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital edema (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 5 (5) | 4 (9) | 2 (6)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (3) | 1 (1) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 2 (4) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 4 (8) | 3 (3) | 0 (0)
Hematoma (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphedema (Vascular disorders) | 0 (0) | 1 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Vascular disorders - Other, specify (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 1 (4) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 5 (9) | 2 (3) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (2) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT04151667/Prot_SAP_000.pdf